CLINICAL TRIAL: NCT03334942
Title: Addressing Community Violence-related Traumatic Stress Symptoms in Children
Brief Title: Addressing Traumatic Stress Symptoms in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Drexel University (Other); University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17-013839; R01HD087406-01A1 (NIH)
Record Dates: First submitted 2017-10-13; First posted 2017-11-07 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Violence, Non-accidental; Posttraumatic Stress Disorder; Parent-Child Relations; Assault; Youth
Keywords: youth; parents; posttraumatic stress; violence; violent injuries
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Research assistants (RAs) will perform eligibility screening in the CHOP ED or Trauma Unit on potentially eligible youth and their caregivers who present for care following an assault-related injury. For individuals discharged before being screened, RAs will phone them within 14 days of discharge for screening. Consented youth and caregivers will complete baseline study assessments followed by random assignment to either the intervention [Violence Intervention Program (VIP) with Child and Family Traumatic Stress Intervention (CFTSI)] or control (VIP-only) conditions. VIP is the standard of care provided to assault injured youth treated in the CHOP ED or Trauma Unit. The study coordinator or VIP staff member will notify youth of their assigned condition. CFTSI clinicians will schedule intervention sessions with the families in community-based mental health centers. RAs will be blinded to participant condition and administer baseline and follow-up assessments to all participants.
Who Masked: Outcomes Assessor
Masking Description: Only the study coordinator and VIP staff members will be aware of a participant's randomization assignment. The study research assistants (RAs), who will be responsible for administering baseline, 4-month, and 10-month assessments will be blinded to the participant's study condition throughout the duration of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CFTSI (Experimental): Youth and caregivers randomized to the Violence Intervention Program (VIP) and Child and Family Traumatic Stress Intervention (CFTSI) arm will receive 5 to 8 CFTSI sessions with a trained clinician and be enrolled in VIP. VIP is the standard clinical service offered to assault injured patients treated in the CHOP ED. Participants in this arm will also complete follow-up assessments approximately 4 and 10 months following the ED visit.
  Interventions: Behavioral: Child and Family Traumatic Stress Intervention
- Violence Intervention Program (No Intervention): Youth and caregivers randomized to the VIP-only condition will complete a baseline assessment prior to randomization and then be enrolled in the Violence Intervention Program (VIP). VIP is the standard clinical service offered to assault injured patients treated in the CHOP ED. Participants in this arm will also complete follow-up assessments approximately 4 and 10 months following the ED visit.

INTERVENTIONS:
Behavioral: Child and Family Traumatic Stress Intervention — The Child and Family Traumatic Stress Intervention (CFTSI) is a 5-8 session intervention, initiated within 60 days of trauma exposure for youth reporting acute PTSS. CFTSI is designed for children age 7 and older, and requires the involvement of a caregiver who knows the child well enough to report changes in the child's behavior and symptoms. CFTSI targets modifiable risk and protective factors during the early post-trauma period to promote recovery and reduce PTSS via caregiver-child communication and cognitive and emotional processing. CFTSI uses skill modules (e.g., sleep disturbance, intrusive thoughts, anxiety) to teach effective strategies to decrease a child's PTSS. Coping and communication skills are taught and practiced in caregiver-child sessions and in the home.
  Other Names: CFTSI
  Arms: CFTSI

SUMMARY:
The objective of this study is to evaluate the effectiveness of the Child and Family Traumatic Stress Intervention (CFTSI), provided soon after a violent traumatic event, in producing significant and sustained reduction in PTSS among assault injured youth.

DETAILED DESCRIPTION:
Interventions to target modifiable risk and protective factors during the early post-trauma period may promote recovery and reduce posttraumatic stress symptoms (PTSS) following violent injury by facilitating cognitive and emotional processing of trauma reactions, increasing coping capacity, and providing emotional support.

Investigators seek to evaluate the effectiveness of the Child and Family Traumatic Stress Intervention (CFTSI), provided soon after a violent traumatic event, in producing significant and sustained reduction in PTSS among assault injured youth.

Participants will be recruited from Children's Hospital of Philadelphia (CHOP) emergency department (ED) or Trauma Unit following interpersonal assault. Investigators seek to enroll 110 participants from CHOP. Participants must reside in Philadelphia County with a caregiver for at least the last six months, be 8 to 18 years of age (inclusive), have been received for an injury resulting from a qualifying interpersonal assault, and both child and caregiver must be able to speak English. Youth must have a Child Post-traumatic stress disorder (PTSD) Symptom Scale (CPSS) score > or = 11 during study screening.The Child and Family Traumatic Stress Intervention (CFTSI) is the study intervention. The primary outcome measure is youth-reported PTSS at 4 and 10 months.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for youth participants

  1. Males or females age 8 to 18 years (inclusive)
  2. Received treatment in the CHOP ED or trauma unit for an injury resulting from a qualifying interpersonal assault
  3. Child must be able to speak English well enough to participate in study activities
  4. Child must reside in Philadelphia County (191xx zip code)
  5. Identifies a consistent caregiver for at least the past 6 months. This may include a parent, legal guardian, or another adult (e.g. grandparent, adult sibling, aunt/uncle, etc.).
  6. Child PTSD Symptom Scale (CPSS) score > or = 11 in ED or on screening telephone call
  7. Parental/guardian permission (informed consent) and child assent
* Inclusion criteria for adult participants

  1. Parent, legal guardian, or other caregiver of an eligible youth participant. Other caregivers may include non-legal guardians who meet all other study eligibility requirements and have approval of the participating child's parent/legal guardian to participate in study activities.
  2. Adult must be able to speak English well enough to participate in study activities
  3. Adult is youth's consistent caregiver for at least the past 6 months
  4. Provide permission (informed consent) to participate in study activities. When a caregiver who is a non-legal guardian is identified to be primary caregiver and meet all other eligibility requirements, parental consent will be obtained for child participation in addition to non-legal guardian consent for self-participation.

Exclusion Criteria:

* Exclusion criteria for youth participants

  1. Age younger than 8 or older than 18 years
  2. Youth who is non-English speaking or for other reasons is unable to understand and answer study questions and participate in study activities
  3. Youth hospitalized for greater than 14 days (unable to achieve timely study enrollment)
  4. No long-term (< 6 months) caregiver
  5. Index injury in the ED due to family violence (assaulted by a parent, sibling, or other family/household member), sexual assault, or fights with police, security, or school personnel
  6. In residential placement at time of ED visit
  7. Parent or legal guardian unable to provide consent for youth participation.
* Exclusion criteria for adult participants

  1. Not a primary or consistent caregiver for eligible youth for at least 6 months
  2. Adult who is non-English speaking or for other reasons is unable to understand and answer study questions and participate in study activities
  3. Unable or unwilling to participate in CFTSI

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 132 (Actual)
Dates: Start 2017-11-02 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Child PTSD Symptom Scale (CPSS-5) score from baseline to 4 months post-ED visit. | 4 months
  Assesses the severity of posttraumatic stress symptoms in youth ages 8 to 18 years old. Items correspond to DSM-5 PTSD symptom criteria. Symptom items are rated on a Likert-type scale (0-1-2-3-4) corresponding to "not at all" to "6 or more times a week/almost always." The CPSS yields a symptom severity score (sum of responses) and can be scored for possible PTSD diagnosis. Possible CPSS-5 scores range from 0 to 80. Based on the current evidence regarding screening for PTSD risk, we will employ a screening cut-off (greater than or equal to 11) on the summed CPSS severity score from 20 symptom items, indicating moderate PTSS.

SECONDARY OUTCOMES:
Change in Revised Children's Anxiety and Depression Scale (RCADS) short form score from baseline to 4 months post-ED visit | 4 months
  Items assess a youth's self-reported anxiety and depression. Response options range from "never" to "always". Item responses are summed to create an RCADS total score with higher scores indicating greater frequency of anxiety and low mood. Possible scores on the short form range from 0 to 75.
Change in Revised Children's Anxiety and Depression Scale (RCADS) short form score from baseline to 10 months post-ED visit | 10 months
  Items assess a youth's self-reported anxiety and depression. Response options range from "never" to "always". Item responses are summed to create an RCADS total score with higher scores indicating greater frequency of anxiety and low mood. Possible scores on the short form range from 0 to 75.
Change in self-reported substance use as assessed by Behavioral Health Screen (BHS) items from baseline to 4 months post-ED visit | 4 months
  Assesses use of alcohol and illicit drugs in participants 12 years of age and older.
Change in self-reported substance use as assessed by Behavioral Health Screen (BHS) items from baseline to 10 months post-ED visit | 10 months
  Assesses use of alcohol and illicit drugs in participants 12 years of age and older.
Change in Strengths and Difficulties Questionnaire-Child and Parent Report (SDQ & SDQ-P) from baseline to 4 months post-ED visit | 4 months
  The SDQ and SDQ-P assess externalizing and internalizing problem areas (conduct problems, hyperactivity/inattention, emotional symptoms, peer problems) as well as pro-social behavior in youth. The measure has age-tailored parent- and self-report versions, with two questions assessing intervention change. Items are scored as "not true", "somewhat true", or "certainly true." The first four problem subscales (emotional symptoms, conduct problems, hyperactivity-inattention, peer problems) are summed to create a Total Difficulties scale score ranging from 0 to 40. Higher scores on the difficulties subscales and Total Difficulties scale correspond to higher levels of difficulty. Higher scores on the prosocial behavior scale indicate higher levels of strengths.
Change in Strengths and Difficulties Questionnaire-Child and Parent Report (SDQ & SDQ-P) from baseline to 10 months post-ED visit | 10 months
  The SDQ and SDQ-P assess externalizing and internalizing problem areas (conduct problems, hyperactivity/inattention, emotional symptoms, peer problems) as well as pro-social behavior in youth. The measure has age-tailored parent- and self-report versions, with two questions assessing intervention change. Items are scored as "not true", "somewhat true", or "certainly true." The first four problem subscales (emotional symptoms, conduct problems, hyperactivity-inattention, peer problems) are summed to create a Total Difficulties scale score ranging from 0 to 40. Higher scores on the difficulties subscales and Total Difficulties scale correspond to higher levels of difficulty. Higher scores on the prosocial behavior scale indicate higher levels of strengths.
Change in Child PTSD Symptom Scale (CPSS-5) score from baseline to 10 months post-ED visit. | 10 months
  Assesses the severity of posttraumatic stress symptoms in youth ages 8 to 18 years old. Items correspond to DSM-5 PTSD symptom criteria. Symptom items are rated on a Likert-type scale (0-1-2-3-4) corresponding to "not at all" to "6 or more times a week/almost always." The CPSS yields a symptom severity score (sum of responses) and can be scored for possible PTSD diagnosis. Possible CPSS-5 scores range from 0 to 80. Based on the current evidence regarding screening for PTSD risk, we will employ a screening cut-off (greater than or equal to 11) on the summed CPSS severity score from 20 symptom items, indicating moderate PTSS.

CONTACTS AND LOCATIONS:
Overall Officials: Joel Fein, MD, MPH, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No